CLINICAL TRIAL: NCT03696433
Title: Visualizing Vascular Mechanisms of Salt Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rachelle Crescenzi, Research Instructor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 181610
Record Dates: First submitted 2018-09-25; First posted 2018-10-04 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Cardiovascular Risk Factor; Salt; Excess
Keywords: salt sensitive, blood pressure, obesity, magnetic resonance imaging
MeSH Terms: conditions — Obesity | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low- then high-salt diet (Experimental): 10 subjects will be enrolled and each will undergo study procedures at 4 separate visits. Subjects will be randomly assigned to this study arm, differing in the order of low and high salt diets. After a baseline visit to include a noninvasive MRI scan, the subject will begin this study diet: low-salt diet, then washout consisting of the subject's typical diet, then high-salt diet. Each dietary or washout period lasts for 7 days, and study visits will occur after each period.
  Interventions: Dietary Supplement: Low-salt diet; Dietary Supplement: High-salt diet
- High- then low-salt diet (Experimental): 10 subjects will be enrolled and each will undergo study procedures at 4 separate visits. Subjects will be randomly assigned to this study arm, differing in the order of low and high salt diets. After a baseline visit to include a noninvasive MRI scan, the subject will begin this study diet: high-salt diet, then washout consisting of the subject's typical diet, then low-salt diet. Each dietary or washout period lasts for 7 days, and study visits will occur after each period.
  Interventions: Dietary Supplement: Low-salt diet; Dietary Supplement: High-salt diet

INTERVENTIONS:
Dietary Supplement: Low-salt diet — The low-salt diet (7 days) will consist of meals, snacks and water provided by Vanderbilt's metabolic kitchen.
Dietary Supplement: High-salt diet — The high-salt diet (7 days) consists of each subject's typical diet, supplemented each day with 2 bullion broth packets, which will be provided to the subject by the study staff.

SUMMARY:
This study aims to assess the salt sensitive blood pressure response to dietary salt load compared with radiological markers of salt handling.

DETAILED DESCRIPTION:
Hypertension is a major cause of heart disease, heart failure, and stroke. Hypertension, or high blood pressure, affects people differently and is related to the body's ability to maintain healthy circulation of salt. Some individuals may be affected by salt sensitive blood pressure (SSBP), when their blood pressure changes in response to dietary salt load. SSBP is a prevalent, independent risk factor for developing cardiovascular disease that preferentially affects black individuals. Current methods to assess SSBP require dietary salt loading over the course of days to weeks, and measurement of blood pressure following high salt diet and low salt diet. Such lengthy protocols are not feasible in a clinical setting to evaluate this risk factor for cardiovascular disease, and more importantly, these procedures provide incomplete information about mechanisms of salt sensitivity.

Our knowledge regarding salt handling in the body is limited. While renal dysfunction is partly responsible for SSBP, recent research points to the role of lymphatic vascular clearance in regulating tissue salt storage and blood pressure control. To better understand these mechanisms in vivo, we have recently developed a noninvasive magnetic resonance (MR) lymphangiography method sensitive to lymphatic vasculature, and applied standardized MR protocols for measuring tissue sodium and fat storage in adults with impaired lymphatic clearance. We found evidence of lymph stasis and tissue salt deposition that correlated with local subcutaneous fat volume. Here, we will test whether similar lymphatic pathways are impaired in persons with SSBP, leading to tissue salt and fat storage, in comparison to the involvement of renal dysfunction in SSBP tissue profiles.

The aims of this study are to improve our understanding of vascular mechanisms of human salt storage, and to provide standardized radiologic biomarkers sensitive to the SSBP phenotype. This study will test the primary hypothesis that the SSBP response is correlated with baseline tissue sodium storage, and elevated in persons with salt sensitivity. Secondary hypotheses will address whether the SSBP response is related to fat storage, lymphatic vascular function, renal vascular function, and impaired target organ responses to salt loading, including decreased urinary sodium excretion, and less suppression of plasma renin and serum aldosterone.

ELIGIBILITY:
Inclusion Criteria:

* Identification as black race
* Age between 18 and 55 years
* Body mass index between 25 and <35 kg/m2
* Normotensive or pre-hypertensive
* Willing to adhere to study diets
* Able to provide informed consent and communicate with study personnel

Exclusion Criteria:

* Prevalent cardiovascular disease or use of medications for cardiovascular disease
* Current or prior history of hypertension or use of blood pressure lowering medications
* Current or prior history of diabetes mellitus or use of anti-diabetic medications
* Prevalent renal disease (eGFR < 60 ml/min/1.73m2), abnormal serum sodium or potassium
* Current or prior smoker
* Current pregnancy, or use of hormone replacement therapy or oral contraceptive
* Current steroid use
* Contraindications to MRI
* Active infection or open wounds on the top of the feet or hands

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle Crescenzi, PhD, Principal Investigator — Department of Radiology, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Crescenzi R, Marton A, Donahue PMC, Mahany HB, Lants SK, Wang P, Beckman JA, Donahue MJ, Titze J. Tissue Sodium Content is Elevated in the Skin and Subcutaneous Adipose Tissue in Women with Lipedema. Obesity (Silver Spring). 2018 Feb;26(2):310-317. doi: 10.1002/oby.22090. Epub 2017 Dec 27. PMID 29280322
- [Background] Crescenzi R, Donahue PMC, Hartley KG, Desai AA, Scott AO, Braxton V, Mahany H, Lants SK, Donahue MJ. Lymphedema evaluation using noninvasive 3T MR lymphangiography. J Magn Reson Imaging. 2017 Nov;46(5):1349-1360. doi: 10.1002/jmri.25670. Epub 2017 Feb 28. PMID 28245075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Black men and women 18-55 years old with BMI 25 to <35 kg/m2 with BP< 140/90 mmHg at screening were recruited as long as they had not used medications for cardiovascular disease, a history of hypertension or diabetes, use of blood pressure or anti-diabetic medications, prevalent renal disease, abnormal serum sodium or potassium. As well as not being a current or prior smoker, pregnant, using hormone replacement therapy, oral contraceptives, or steroids, or had contraindications to MRI.
Pre-assignment Details: Participants went through a screening process with a physician to determine health and study qualifications. Once screening was complete, participants were assigned to either low-salt or high-salt diet study arm.
Period: Overall Study
Arm/Group | Low- Then High-salt Diet | High- Then Low-salt Diet
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low- Then High-salt Diet | High- Then Low-salt Diet | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.4 [19 to 37] | 28.1 [20 to 47] | 26.8 [19 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19
Tissue Sodium Content of the Leg [Mean (Standard Deviation); unit: mmol/L] — Measured by standardized sodium 23Na 3.0T MRI in the leg at the widest part of the calf. Population: Tissue sodium content was not obtained in some participants in the low-then-high-salt diet group.
  mmol/L
    number analyzed (Participants) | 6 | 10 | 16
    (all) | 14.84 (1.50) | 14.33 (3.06) | 14.60 (2.61)

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure Following High-salt Diet and Low-salt Diet
Description: Mean arterial pressure following high-salt diet and low-salt diet
Time Frame: Following completion of all dietary supplements and washout, in no less than 21 days.
Population: All Subjects received both a low salt diet and high salt diet. Data reported reflects measure of mean arterial blood pressure following high-salt diet and low-salt diet.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Low Salt Diet: Low-salt diet: The low-salt diet (7 days) will consist of meals, snacks and water provided by Vanderbilt's metabolic kitchen.
- High Salt Diet: High-salt diet: The high-salt diet (7 days) consists of each subject's typical diet, supplemented each day with 2 bullion broth packets, which will be provided to the subject by the study staff.
Arm/Group | Low Salt Diet | High Salt Diet
Number analyzed (Participants) | 19 | 19
mmHg | 83.3 (21.4) | 89.5 (9.55)

ADVERSE EVENTS:
Time Frame: Baseline up to 8 weeks
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion.
Arm/Group | Low Salt Diet | High Salt Diet
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Salt Diet (N=19) | High Salt Diet (N=19)
episode of syncope (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT03696433/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03696433/SAP_001.pdf